CLINICAL TRIAL: NCT06647017
Title: Delivering Transcutaneous Auricular Neurostimulation to Reduce Blood Loss During Dialysis AV Graft Placement Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Surgical Vascular (Industry)
Collaborators: Spark Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1983231
Record Dates: First submitted 2024-10-04; First posted 2024-10-17 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Blood Loss, Surgical
Keywords: auricular neurostimulation; vagus nerve stimulation; transcutaneous; blood loss; transcutaneous auricular neurostimulation; tAN
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants and investigator will be blind to participant treatment group assignment. Only the research coordinator will know treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tAN + standard of care (Experimental): Participants randomized to the active group will have an earpiece applied and receive 30 minutes of active tAN therapy immediately prior to the dialysis port placement procedure. When the 30-minute tAN session is complete, the system will be turned off, unplugged, and the earpiece will be removed.
  Interventions: Device: Volta tAN System
- Sham tAN + standard of care (Sham Comparator): Participants randomized to the sham group will have an earpiece applied, but stimulation will not be turned on. These participants will receive 30 minutes of sham tAN therapy immediately prior to the dialysis port placement procedure. When the 30-minute tAN session is complete, the system will be turned off, unplugged, and the earpiece will be removed.
  Interventions: Device: SHAM Volta tAN System

INTERVENTIONS:
Device: Volta tAN System — Transcutaneous auricular neurostimulation (tAN)
  Other Names: Sparrow Ascent
  Arms: Active tAN + standard of care
Device: SHAM Volta tAN System — Participants randomized to the sham group will have an earpiece applied, but stimulation will not be turned on.
  Other Names: Sparrow Ascent
  Arms: Sham tAN + standard of care

SUMMARY:
The objective of this study is to determine if tAN therapy can reduce the volume of blood lost during dialysis AV graft placement procedures.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, sham-controlled, single-center, pilot clinical trial in which adults undergoing dialysis port placement procedures will be randomized 1:1 into one of two treatment groups:

Group 1: Active tAN + standard of care Group 2: Sham tAN + standard of care

Participants will receive 30 minutes of active or sham tAN immediately prior to the dialysis port placement procedure. Blood loss and blood markers will be measured before and during the procedure to measure the effect of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is undergoing a dialysis port placement procedure using synthetic graft
* Participant is between 18 and 75 years of age
* Participant is English proficient
* Participant is able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

* Participant has a BMI ≥ 40
* Participant is currently taking a platelet inhibitor medication
* Participant has a history of epileptic seizures
* Participant has a history of neurological diseases or traumatic brain injury
* Participant has presence of devices, e.g., pacemakers, cochlear prosthesis, neurostimulators
* Participant has abnormal ear anatomy or ear infection present
* Person of childbearing age, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study
* Person who is pregnant or lactating
* Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean Total Blood Loss | Throughout procedure
  Comparison of mean total quantified blood loss in active tAN versus sham tAN groups.

SECONDARY OUTCOMES:
Surgery Time | First incision to incision closure
  Surgery time measured as total time from first incision to incision closure in active tAN versus sham tAN groups.
Time to Hemostasis | From end of AV graft placement to beginning of surgical site closure
  Comparison of mean time to hemostasis in active tAN versus sham tAN groups.

OTHER OUTCOMES:
Hemostatic Agent Use | During surgery
  Proportion of participants requiring hemostatic agents
Duration of time between completing graft placement and application/administration of hemostatic agent | During surgery
  Duration of time between completing graft placement and application/administration of hemostatic agent
Proportion of participants achieving hemostasis in <10 minutes | During surgery
  Proportion of participants achieving hemostasis in <10 minutes
Blood Assay Results | Prior to device placement, during surgery, and at end of surgery
  Blood urea nitrogen (BUN) levels, platelet count, hematocrit, and activated clotting time (ACT)
Treatment-Related Adverse Events (Safety) | Thorough study completion, an average of 4 hours
  The proportion of participants who experience one or more treatment-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- University Surgical Vascular, Watkinsville, Georgia, United States